CLINICAL TRIAL: NCT01264900
Title: Cognitive Behavioral Aggression Treatment: Effects on Brain and Behavior
Brief Title: Cognitive Behavioral Aggression Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Principal Investigator, Michael McCloskey, Associate Professor, Temple University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH086525
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Aggression
Keywords: Psychotherapy; Cognitive Behavioral Therapy; Aggression; fMRI; Behavioral Intervention
MeSH Terms: conditions — Aggression | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Twelve weekly 50-minute sessions of individual cognitive behavioral aggression treatment
  Interventions: Behavioral: Psychotherapy
- Supportive Psychotherapy (Active Comparator): Twelve weekly 50-minute sessions of individual supportive (client-centered) psychotherapy
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — Twelve weekly 50-minute sessions of individual cognitive behavioral aggression treatment or supportive psychotherapy
  Other Names: CBT

SUMMARY:
Aggressive behavior is a leading worldwide public health problem. Despite this, relatively little is known about how to best treat individuals who are highly angry and aggressive. A rich literature suggests that aggression is associated with a tendency to interpret situations as threatening or hostile even when they are not. This process is governed by a prefrontal-limbic circuit in the brain. A goal of cognitive behavioral therapy is to reduce these kinds of hostile biases. Preliminary data by the PI suggests a 12- session cognitive behavioral aggression treatment (CBAT) may help reduce aggressive behavior and underlying hostile biases associated with affective aggression. To assess the efficacy of this treatment, 120 adults with high levels of anger and aggression will receive 12 sessions of either CBAT or supportive psychotherapy. All subjects will monitor their anger and aggressive behavior throughout the treatment electronic diaries. Subjects will also complete questionnaires and computer tasks to assess anger, hostile biases and related processes 1-week before treatment begins, and again 1-week, 6-months and 1-year after treatment ends. In addition, to understand the effects of CBAT on the brain, subjects will have their brains scanned (functional Magnetic Resonance Imaging) while they look at emotional pictures and complete computer tasks. The brain scans will occur once before treatment starts and once after treatment ends.

Our hypotheses are:

1. CBAT will reduce anger, aggression and hostile biases more than supportive therapy.
2. CBAT will decrease limbic activation and increase prefrontal activation to emotional pictures more than supportive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Three or more acts of physical aggression (assault / property destruction) in past six months
* Aggression related distress and/or impairment
* Meets Criteria for Intermittent Explosive Disorder

Exclusion Criteria:

* Life History of DSM-IV Axis Bipolar disorder, Schizophrenia, Delusional disorder, Organic disorder, or Mental Retardation
* Current DSM-IV Major Depressive Episode, Alcohol Dependence or other Drug Dependence
* Current (past month) psychotropic medication use
* Current severe suicidal or homicidal ideation necessitating immediate medical intervention
* Current pregnancy or nursing, or existence of any medical condition that would deem the subject ineligible to undergo an fMRI (e.g., metal pins)
* Two consecutive positive Expired Breathalyzer Alcohol or Urine Drug toxicological screens
* Unable or unwilling to cooperate with study protocol (e.g., keep appointments, complete rating forms, read and understand informed consent).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Aggressive Acts | Pre-intervention thru 1 year post-intervention
  Aggressive acts will be measured using electronic diaries and clinical interview

SECONDARY OUTCOMES:
Brain activation to emotional stimuli | 14 weeks
  Brain response (as measured by fMRI)to emotional expressions and pictures

CONTACTS AND LOCATIONS:
Overall Officials: Michael S McCloskey, Ph.D, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] McCloskey MS, Noblett KL, Deffenbacher JL, Gollan JK, Coccaro EF. Cognitive-behavioral therapy for intermittent explosive disorder: a pilot randomized clinical trial. J Consult Clin Psychol. 2008 Oct;76(5):876-86. doi: 10.1037/0022-006X.76.5.876. PMID 18837604